CLINICAL TRIAL: NCT05520190
Title: Acceptability and Feasibility of Cognitive Behavioral Therapy for Treatment-Seeking (CBT-TS) With Deaf Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Aileen Aldalur, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007447
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Mental Health Issue; Alcohol Use Disorder; Depression; Anxiety; Insomnia; Post Traumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Treatment Seeking (CBT-TS)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Treatment Seeking (CBT-TS) — The intervention will consist of 1 - 2 sessions. The first session is approximately 60 - 90 minutes and will be structured in 4 phases 1) subject's history of symptoms and current functioning, 2) their coping methods, 3) modification of treatment beliefs, 4) action planning. The interventionist will provide the subject with a list of resources for seeking treatment.
  All subjects will be offered an optional second session with the interventionist. The second session will consist of a 60-minute appointment focused on providing practical assistance to identify available treatment options in the subject's area, scheduling treatment sessions, and problem-solving barriers to treatment.

SUMMARY:
The current study aims to assess the acceptability and feasibility of an adapted version of Cognitive Behavioral Therapy for Treatment Seeking (CBT-TS) for use with signing Deaf adults. This is a Stage 1A intervention refinement study consisting of a single-arm open pilot trial. Thirty Deaf adults with clinically significant symptoms of alcohol use disorder (AUD), post-traumatic stress disorder (PTSD), depression, anxiety, and/or insomnia, who are not currently engaged in treatment will be recruited from across the United States. All subjects will complete a baseline assessment of their behavioral health symptoms, perceptions towards treatment, and intent to seek treatment prior to engaging in the adapted CBT-TS intervention. The primary clinical outcome, assessed at one-month follow-up, will be whether subjects scheduled professional treatment. Secondary outcomes include changes in subjects' perceptions towards treatment, intentions to seek treatment, and symptom severity from baseline. During the one-month, follow-up assessment subjects will also complete a client satisfaction survey and open-ended questions to provide feedback about the CBT-TS intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* self-identify as Deaf or hard-of-hearing (any degree of hearing loss)
* primary method of communication is ASL or PSE
* positive screen for one or more behavioral health disorders including: AUD (AUDIT > 16 and alcohol use in the past 30 days exceeds the limit for low-risk drinking established by the NIAAA), PTSD (PCL-5 > 31), depression (PHQ-9 > 10), anxiety (GAD-7 > 10), or insomnia (ISI > 15)
* no current behavioral health treatment per standardized self-report
* access to video chat technology with internet and webcam.

Exclusion Criteria:

* unable to communicate with the researcher in ASL or PSE
* current alcohol withdrawal necessitating medical evaluation
* current psychiatric impairment necessitating emergency services or inpatient admission (i.e., imminent danger of harm to self or others)
* unable to comprehend the nature of the study
* currently receiving behavioral health treatment for their symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aileen Aldalur, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 42
Completed | 33
Not Completed | 9
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 2 participants were lost to follow-up before completing the baseline assessment.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.33 (13.99)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 26
  Male | 13
  Nonbinary | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 27
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Schedule Professional Treatment
Description: We will use a validated treatment utilization survey that will assess subjects' use of 12 treatment services, their reasons for seeking/not seeking treatment, and any barriers they experienced through a series of structured questions. Treatment-seeking will be coded as a binary variable representing those who scheduled or attended any professional treatment service and those who did not.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 33
Participants | 8

2. Primary Outcome: Mean Change in Attitudes About Treatment
Description: The Deaf Perceptions About Services Scale (PASS-D) Attitude scale. The Attitude scale contains 4 items assessing individuals' attitudes about behavioral health treatment. The items are rated on a Likert scale ranging from 1 - 7. Scores are averaged across the items for a total score of 1 - 7 with higher scores indicating more favorable attitudes about treatment.
Time Frame: baseline to 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline Attitude | 4.93 (1.26)
  1-month Attitude | 5.40 (1.25)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = -0.47 — Baseline Attitude score - 1-month Attitude score / SD of average change

3. Primary Outcome: Mean Change in Subjective Norm About Treatment
Description: The Deaf Perceptions About Services Scale (PASS-D) Subjective Norm scale. The Subjective Norm scale contains 3 items assessing individuals' perceptions of the subjective norm in their community about behavioral health treatment. The items are rated on a Likert scale ranging from 1-7. Scores are averaged across the items for a total score of 1 - 7 with higher scores indicating more favorable perceptions about treatment.
Time Frame: baseline to 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline Norms | 5.18 (1.39)
  1-month Norms | 5.51 (0.88)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = -0.23 — Baseline Norm score - 1-month Norm score / SD of average change

4. Primary Outcome: Mean Change in Perceived Behavioral Control About Seeking Treatment
Description: The Deaf Perceptions About Services Scale (PASS-D) Perceived Behavioral Control scale. The Perceived Behavioral Control scale contains 3 items assessing individuals' perceived behavioral control to seek behavioral health treatment. The items are rated on a Likert scale ranging from 1 - 7. Scores are averaged across the items for a total score of 1 - 7 with higher scores indicating more perceived behavioral control to seek treatment.
Time Frame: baseline to 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline Perceived Behavioral Control | 6.10 (1.01)
  1-month Perceived Behavioral Control | 6.14 (1.15)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = -0.03 — Baseline Perceived Behavioral Control score - 1-month Perceived Behavioral Control score / SD of average change

5. Primary Outcome: Mean Change in Intention to Seek Treatment
Description: The D-PASS will be administered pre-and-post-treatment to collect information about subjects' intention to seek treatment. The scale ranges from 3 to 21 with higher scores indicating more favorable attitudes.
Time Frame: baseline to 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline Intention | 4.62 (1.79)
  1-month Intention | 4.92 (2.06)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = -0.16 — Baseline Intention score - 1-month Intention score / SD of average change

6. Post Hoc Outcome: Mean Change in Past Month Drinks Per Day
Description: The National Survey on Drug Use and Health (NSDUH) 30-day alcohol consumption: drinks per day question will assess the average number of drinks per day an individual consumed on days with alcohol consumption in the past month.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | All Participants
Number analyzed (Participants) | 33
drinks per day
  Baseline drinks per day | 1.42 (1.95)
  1-month drinks per day | 0.88 (1.58)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 0.35 — Baseline drinks per day - 1-month drinks per day / avg change in drinks per day

7. Post Hoc Outcome: Mean Change in Past Month Alcohol Drinking Days
Description: The National Survey on Drug Use and Health (NSDUH) 30-day alcohol consumption: drinking days question will assess the number of days the individual consumed alcohol in the past month.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 33
days
  Baseline drinking days | 4.06 (7.08)
  1-month drinking days | 2.64 (0.88)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 0.35 — Baseline drinking days - 1-month drinking days / SD of avg change in drinking days

8. Post Hoc Outcome: Mean Change in Past Month Binge Drinking Days
Description: The National Survey on Drug Use and Health (NSDUH) 30-day alcohol consumption: binge drinking days question will assess the number of days with binge drinking episodes in the past month.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 33
days
  Baseline binge drinking days | 1.15 (4.39)
  1-month binge drinking days | 0.24 (1.39)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 0.30 — Baseline binge drinking days - 1-month binge drinking days / avg change in binge drinking days

9. Post Hoc Outcome: Depression
Description: The Patient Health Questionnaire - 9 (PHQ-9). The PHQ-9 is a 9-item self-report scale assessing the presence and severity of symptoms of depression. Each item is rated on a Likert scale of 0 (not at all) to 3 (nearly every day). Total scores range from 0 - 27 with higher scores indicating more severe depression.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline depression | 13.39 (6.17)
  1-month depression | 7.88 (5.73)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 1.23 — Baseline depression - 1-month depression / SD of avg change in depression

10. Post Hoc Outcome: Anxiety
Description: Generalized Anxiety Scale- 7 (GAD-7). The GAD-7 is a self-report measure of the presence and severity of anxiety symptoms. It contains 7 items rated on a Likert scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0 - 21 with higher scores indicating more severe anxiety symptoms.
Time Frame: Baseline to 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline anxiety | 11.64 (5.61)
  1-month anxiety | 7.27 (1.06)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 1.06 — Baseline anxiety - 1-month anxiety / SD avg change in anxiety

11. Post Hoc Outcome: Post-traumatic Stress Disorder
Description: PTSD Checklist for DSM-5 (PCL-5). The PCL-5 is a 20-item self-report measure of that assesses the 20 DSM-5 symptoms of PTSD. Items are rated on a Likert scale ranging from 0 (not at all) to 4 (Extremely). Total scores range from 0 to 80 with higher scores indicating more severe symptoms of PTSD.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline PTSD | 36.48 (18.06)
  1-month PTSD | 21.94 (16.06)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 0.90 — Baseline PTSD - 1-month PTSd / SD avg change in PTSD

12. Post Hoc Outcome: Insomnia
Description: Insomnia Severity Index (ISI). The ISI is a self-report measure of sleep problems. The scale contains 7 items rated on a Likert scale ranging from 0 to 4. Total scores range from 0 - 28 with higher scores indicating more severe sleep disturbance.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline insomnia | 15.36 (5.99)
  1-month insomnia | 11.93 (7.01)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 0.60 — Baseline insomnia - 1-month insomnia / SD avg change in insomnia

13. Post Hoc Outcome: Mean Change in Symptoms of Alcohol Use Disorder
Description: The Alcohol Use Disorder Identification Test (AUDIT) is a 10-item screening tool that assesses alcohol consumption, drinking behaviors, and alcohol-related problems. Scores range from 0 - 40 with greater scores indicating higher levels of consumption and alcohol-related problems.
Time Frame: baseline to 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline Alcohol Screen | 4.61 (5.49)
  1-month Alcohol Screen | 2.39 (4.34)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = 0.58 — Baseline Alcohol Screen - 1-month Alcohol Screen / SD avg change

14. Post Hoc Outcome: Mean Change in Behavioral Beliefs About Treatment
Description: The Deaf Perceptions About Services Scale (PASS-D) Behavioral beliefs scale. The Behavioral Beliefs Scale contains 10 items that assess individuals' behavioral beliefs about seeking behavioral health treatment. The items are rated on a Likert scale ranging from 1 - 7. Scores are averaged across the items for a total score of 1 - 7 with higher scores indicating more positive behavioral beliefs about seeking treatment.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline behavioral beliefs | 4.88 (0.99)
  1-month behavioral beliefs | 5.31 (0.70)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = -0.39 — Baseline behavioral beliefs - 1-month behavioral beliefs / avg change in behavioral beliefs

15. Post Hoc Outcome: Mean Change in Normative Beliefs About Treatment
Description: The Deaf Perceptions About Services Scale (PASS-D) Normative Beliefs scale. The Normative Beliefs Scale contains 7 items that assess individuals' normative beliefs about behavioral health treatment. The items are rated on a Likert scale ranging from 1 - 7. Scores are averaged across the items for a total score of 1 - 7 with higher scores indicating more positive normative beliefs about treatment.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline normative beliefs | 5.13 (1.00)
  1-month normative beliefs | 5.68 (0.90)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = -0.62 — Baseline normative beliefs - 1-month normative beliefs / SD avg change in normative beliefs

16. Post Hoc Outcome: Mean Change in Control Beliefs About Seeking Treatment
Description: The Deaf Perceptions About Services Scale (PASS-D) Control Beliefs scale. The Control Beliefs Scale contains 26 items that assess individuals' control beliefs about seeking behavioral health treatment. The items are rated on a Likert scale ranging from 1 - 7. Scores are averaged across the items for a total score of 1 - 7 with higher scores indicating more positive control beliefs about seeking treatment.
Time Frame: Baseline to 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 33
score on a scale
  Baseline control beliefs | 4.26 (0.71)
  1-month control beliefs | 4.94 (0.93)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; Standardized Response Mean = -0.83 — Baseline control beliefs - 1-month control beliefs / SD avg change in control beliefs

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT05520190/Prot_SAP_000.pdf